CLINICAL TRIAL: NCT05665439
Title: Study on Local Treatment for Patients With Bone Metastases
Brief Title: Local Treatment for Bone Metastases
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai 6th People's Hospital (Other)
Responsible Party: Principal Investigator, Zhao Hui, Principal Investigator, Shanghai 6th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20221201
Record Dates: First submitted 2022-12-17; First posted 2022-12-27 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Bone Metastases
MeSH Terms: interventions — Radiation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- local treatment (Experimental)
  Interventions: Radiation: radiation
- observation (No Intervention)

INTERVENTIONS:
Radiation: radiation — radiation for patients with newly diagnosed bone metastases or patients with bone metastases after vertebroplasty
  Arms: local treatment

SUMMARY:
This study will carry out a prospective randomized controlled study to study the effect of different local treatment on disease control, quality of life, economic cost and even survival period of patients by randomly giving local radiotherapy or observation to patients with newly diagnosed bone metastases or patients with bone metastases after vertebroplasty.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are definitely diagnosed as malignant tumor by pathology or cytology;
2. At least one bone metastasis site;
3. Aged over 18;
4. ECOG：0-1；
5. The pain score is less than 5 or after vertebroplasty within 1 month.

Exclusion Criteria:

1. The expected life span is less than 3 months;
2. Spinal metastatic tumor stability score (SINS) is greater than 7;
3. Spinal cord compression;
4. The patient refused the treatment decision of the integrated team.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 348 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Disease control rate at 1 year | 1 year
  Disease control rate

SECONDARY OUTCOMES:
Progression-Free Survival | 1 year
Overall Survival | 1 year